CLINICAL TRIAL: NCT01471223
Title: Belatacept in Renal Transplantation: Analyses Using Data From the Collaborative Transplant Study (CTS)
Brief Title: Belatacept in Renal Transplantation: Analyses Using Data From the Collaborative Transplant Study
Acronym: CTS
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: IM103-089
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients receiving Belatacept in CTS: Patients receiving a 1st kidney-only transplant at a center participating in the CTS and receiving Belatacept at the time of transplantation
- Patients receiving CNI in CTS: Patients receiving a 1st kidney-only transplant at a center participating in the CTS and receiving CNI at the time of transplantation

SUMMARY:
The purpose of the study is to estimate the incidence rates of Post-transplant Lymphoproliferative Disorder (PTLD), malignancy and hospitalized infections in adult kidney-only transplant recipients treated with Belatacept, and compared the incidences to the incidences in those treated with Calcineurin inhibitor (CNI) based regimens at the time of transplantation.

DETAILED DESCRIPTION:
Time Perspective: Prospective design, Retrospective data collection and analysis

ELIGIBILITY:
Inclusion Criteria:

* 1st kidney only transplant during study, at one of the transplant centers participating in CTS, received Belatacept or a CNI at the time of transplantation

Exclusion Criteria:

* Patients with a history of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing 1st kidney only transplantation, whose transplant centers participate in CTS and who are treated with Belatacept or a CNI based regimen at the time of transplantation
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Incidences of Post-transplant Lymphoproliferative Disorder (PTLD) | 5 years post transplantation
Incidences of hospitalized infections | 2 years post transplantation
Incidences of malignancy | 5 years post transplantation

SECONDARY OUTCOMES:
Incidence rates of PTLD in adult subgroups of Belatacept- vs. CNI-treated, kidney-only transplant recipients defined by donor-recipient Epstein Barr virus (EBV) serostatus and by age groups | Every 6 months and 12 months
Location, mortality, and tumor type of all PTLD cases in adult kidney-only transplant recipients treated with Belatacept vs. CNI-based regimens at the time of transplantation and in subgroups of these transplant recipients | Every 6 months and 12 months
  Subgroups of the transplant recipients defined by donor-recipient EBV serostatus at the time of transplantation
Cumulative incidence of hospitalized infections in adult kidney-only transplant recipients treated with Belatacept vs. CNI-based regimens at the time of transplantation | Every 6 months and 12 months
  Hospitalized infections for the following infection groups:
  1. Bacterial
  2. fungal
  3. Viral
  4. Tuberculosis
  5. Herpes and
  6. Cytomegalovirus (CMV)
Incidence rates of graft rejection in adult kidney-only transplant recipients treated with Belatacept vs. CNI-based regimens at the time of transplantation | Every 6 months and 12 months
Incidence rates of graft failure in adult kidney-only transplant recipients treated with Belatacept vs. CNI-based regimens at the time of transplantation | Every 6 months and 12 months
Mortality rate of composite bacterial, fungal, viral, tuberculosis, herpes, and CMV infections | 2 years post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm